CLINICAL TRIAL: NCT01046630
Title: A Phase I, Multi-centre, Double-blind, Placebo-controlled Parallel Group Study to Assess the pharmacoMRI Effects of AZD6765 in Male and Female Subjects Fulfilling the Criteria for Major Depressive Disorder
Brief Title: Study Where Pharmaco Magnetic Resonance Imaging (MRI) Effects of AZD6765 Will be Compared to Placebo in Depressive Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: University of Manchester (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: D2285C00001
Record Dates: First submitted 2010-01-05; First posted 2010-01-12 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: Phase I; BOLD signal; fMRI; AZD6765; BOLD signal measured by fMRI
MeSH Terms: conditions — Depression | interventions — AZD6765; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): single infusion
  Interventions: Drug: AZD6765
- 2 (Active Comparator): single infusion
  Interventions: Drug: Ketamine
- 3 (Placebo Comparator): single infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6765 — single infusion
  Arms: 1
Drug: Ketamine — single infusion
  Arms: 2
Drug: Placebo — single infusion
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effect of a single dose infusion of AZD 6765 compared with placebo and ketamine on the blood oxygen level dependent signal using fMRI (functional Magnetic Resonance Imaging) in depressed subjects.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis meeting criteria from the DSM-IV by structured clinical interview,major depressive disorder, single episode or recurrent
* Outpatient status at screening and at randomisation

Exclusion Criteria:

* A major depression disorder which has a major impact on the subjects current psychiatric status
* Subjects not allowed to use mood stabilizers, antidepressants or other antipsychotic or psychoactive drugs
* Subjects with lifetime history of schizophrenia, bi-polar, psychosis and psychotic depression

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Measurements of BOLD signal in the brain area BA25 | Day1 (at infusion)

SECONDARY OUTCOMES:
Measurements of symptoms of depression using Montgomery-Asberg Depression Rating Scale and Beck Depression Inventory total score | once during Day -30 to Day -1, twice Day 1 (pre and 4hrs post infusion) [BDI only pre-infusion], once Day 2 (approx 24hrs post infusion), once Day 9-12
Responses on a computer based battery of behavioral tasks | Day2 (approx 24 post infusion)
Pharmacokinetics of AZD6765 | Max 3 times Day1 (pre-infusion, end of infusion, 4 hrs end of infusion), Max once Day2 (approx 24 hrs post infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Deakin, Prof, Principal Investigator — University of Manchester, Neurosciance and Psychiatry Unit, UK; Guy Goodwin, Prof, Principal Investigator — University of Oxford, Departmentof Psychiatry, UK; Malene Jensen, Study Director — AstraZeneca R&D, Södertälje, Sweden
Locations (2):
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Oxford

REFERENCES:
- [Derived] Downey D, Dutta A, McKie S, Dawson GR, Dourish CT, Craig K, Smith MA, McCarthy DJ, Harmer CJ, Goodwin GM, Williams S, Deakin JF. Comparing the actions of lanicemine and ketamine in depression: key role of the anterior cingulate. Eur Neuropsychopharmacol. 2016 Jun;26(6):994-1003. doi: 10.1016/j.euroneuro.2016.03.006. Epub 2016 Apr 28. PMID 27133029
- See also: D2285C00001 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1244&filename=D2285C00001_Clinical_Study_Report_Synopsis.pdf